CLINICAL TRIAL: NCT06723652
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study Evaluating the Efficacy and Safety of SHR-1918 in Patients With Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1918-301
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2024-12

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1918 (Experimental)
  Interventions: Drug: SHR-1918
- SHR-1918 placebo (Placebo Comparator)
  Interventions: Drug: SHR-1918 placebo

INTERVENTIONS:
Drug: SHR-1918 — six administration
  Arms: SHR-1918
Drug: SHR-1918 placebo — SHR-1918 placebo three administration+SHR-1918 three administration
  Arms: SHR-1918 placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study to assess the reduction of low-density lipoprotein cholesterol (LDL-C) by SHR-1918 in patients with homozygous familial hypercholesterolemia (HoFH).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of functional HoFH by either genetic or clinical criteria as defined in the protocol
2. LDL-C ≥2.6mmol/L at the screening visit
3. Body weight ≥40 kg
4. Receiving stable lipid-lowering therapy for at least 28 days before enrollment.

Exclusion Criteria:

1. Treatment with an ANGPTL3 inhibitor within 24 weeks prior before screening
2. Previously diagnosed type 1 diabetes or poorly controlled type 2 diabetes at screening (HbA1c > 8.5%)
3. eGFR <30ml/min/1.73m2 at the screening visit
4. CK >5times ULN at the screening visit

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Percent change in calculated LDL-C from baseline to week 12 | week 12

SECONDARY OUTCOMES:
Change in calculated LDL-C from baseline to week 12 | week 12
Percent change and changer in calculated LDL-C from baseline to week 24 | week 24

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided